CLINICAL TRIAL: NCT06561087
Title: Phase II Randomized, Placebo- Controlled Study of Intralesional Nivolumab for High-risk Oral Premalignant Lesions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0022; NCI-2024-06909 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Premalignant Lesion
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab/Placebo (Experimental): Participants will be screened for LOH and randomly assigned to trial
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Given by injections
  Other Names: BMS-936558, Opdivo

SUMMARY:
To evaluate the antitumor efficacy of intralesional injections of nivolumab in patients with high-risk oral premalignant lesions

DETAILED DESCRIPTION:
Primary Objectives:

To assess the oral cancer free survival following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions

Secondary Objectives:

To describe the objective response rate (ORR) in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions, according to modified World Health Organization (WHO) criteria.

To describe the pathologic complete response (CR) rate in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions.

To describe the major pathologic response rate in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a treatment naïve, biopsy proven, intraoral premalignant lesion visible from oral cavity.
2. Be willing and able to provide written informed consent for the trial. In the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an ICD in their language, will be utilized and completed in accordance with the MDACC "Policy For Consenting Non-English Speaking Participants."
3. Be >/= 18 years of age on day of signing informed consent.
4. Be willing to provide tissue, either archive or from a newly obtained oral biopsy.
5. Have a performance status of 0-2 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined in Table 1
7. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of study therapy through 120 days after the last dose of Nivolumab. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy with potential anti-neoplastic activity or has participated in a study of an investigational agent and received study therapy with potential anti-neoplastic activity within 4 weeks of the first dose of treatment.
2. Has a known history of active TB (Bacillus Tuberculosis)
3. Hypersensitivity to nivolumab or any of its excipients.
4. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 2 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 2 or at baseline) from adverse events due to a previously administered agent.
6. Has a known additional malignancy that is progressing or requires active treatment other than adjuvant hormonal therapy. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin or in situ cervical cancer.
7. Has known history of, or any evidence of active, non-infectious pneumonitis.
8. Has an active infection requiring systemic therapy.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of treatment with nivolumab, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
12. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety and AdverseEevents (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Moran Amit, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org